CLINICAL TRIAL: NCT06857266
Title: Remote Video-Delivered Suturing Education with Smartphones: a Non-Inferiority Randomized Controlled Trial
Brief Title: Remote Video-Delivered Suturing Education with Smartphones
Acronym: REVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 11324
Record Dates: First submitted 2024-11-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-09

CONDITIONS: Surgical Skill Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-person teaching (Active Comparator)
  Interventions: Other: In-Person Feedback
- Live Video Feedback (Experimental)
  Interventions: Other: Live Video-delivered Feedback
- Recorded Video Feedback (Experimental)
  Interventions: Other: Recorded Video-delivered feedback

INTERVENTIONS:
Other: Live Video-delivered Feedback — Feedback is delivered to students through a live video call.
  Arms: Live Video Feedback
Other: In-Person Feedback — In-Person Feedback
  Arms: In-person teaching
Other: Recorded Video-delivered feedback — Feedback is delivered via a personalized recorded video made by the instructor specific to the student's performance.
  Arms: Recorded Video Feedback

SUMMARY:
Medical students were randomized to receive live video- or recorded video-delivered feedback on suturing skills. A non-randomized control group received in-person feedback. Pre- and post-feedback recordings of suturing were evaluated to see if the students receiving video-delivered feedback improved just as much as students receiving in-person feedback.

DETAILED DESCRIPTION:
Medical students were randomized to receive live video- or recorded video-delivered feedback on suturing skills. A non-randomized control group received in-person feedback. Pre- and post-feedback recordings of suturing were evaluated by blinded assessors to determine improvement using the University of Bergen suturing skills assessment tool (UBAT) and Objective Structured Assessment of Technical Skills (OSATS). Study arms were compared to the control arm in a non-inferiority analysis. Participants and feedback providers completed questionnaires regarding feasibility and utility of their feedback modality.

ELIGIBILITY:
Inclusion Criteria:

* First and second year students at McMaster University's Degroote School of Medicine

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in University of Bergen suturing skills Assessment Tool score | At 48 hours after feedback given to student

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada